CLINICAL TRIAL: NCT00878527
Title: Safety and Performance Evaluation of the CircuLite Synergy Pocket Circulatory Assist Device
Brief Title: Safety and Performance Evaluation of CircuLite Synergy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CircuLite CRP-001
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Heart Failure
Keywords: Heart Failure; Partial Circulatory Assist; NYHA Class IIIb; NYHA Class IV; Ventricular Assist Device; VAD
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment with the pump (Experimental): Treatment with the CircuLite Synergy Pocket Circulatory Assist Device
  Interventions: Device: CircuLite Synergy Pocket Circulatory Assist Device

INTERVENTIONS:
Device: CircuLite Synergy Pocket Circulatory Assist Device — Goal of successful implantation and follow-up for at least three months
  Other Names: CircuLite; CircuLite Synergy; CircuLite Micro pump; CircuLite Synergy Partial Circulatory Assist Device

SUMMARY:
The purpose of the study is to demonstrate the safety and functionality of the CircuLite Synergy Pocket Circulatory Assist Device.

DETAILED DESCRIPTION:
The CircuLite Synergy Pocket Circulatory Assist Device is an implantable miniature, mixed-flow blood pump designed o provide partial left ventricular support in patients with advanced heart failure. Treatment for this patient population currently include lifestyle changes, medicines, transcatheter interventions and surgery, including implantation of mechanical ventricular assist devices (VADs); most of the currently available VADs require highly invasive, high-risk surgical procedures to implant due to large device size, and are therefore generally limited to use in patients with terminal heart failure. The Synergy pump is intended for treatment of patients with New York Heart Association (NYHA) Class III and IV heart failure; it is expected that the pump will provide these patients with 2-3 L/min of additional blood flow, giving adequate cardiac support to increase exercise tolerance and improve patients' quality of life. The pump's small size will allow it to be implanted in a less surgically invasive procedure than used with previous VADs, which should result in a reduction of perioperative morbidity. The device wil be implanted in a left atrial to subclavian artery bypass with the pump being located in the infraclavicular fossa like a pacemaker.

ELIGIBILITY:
Inclusion Criteria:

* Maximum tolerable medical therapy including ACE inhibitors and Beta Blockers
* NYHA Class III or IV despite maximal tolerable medical therapy
* Ambulatory (inpatient or outpatient)
* Patients on the heart transplant list (or, not currently listed but otherwise suitable for heart transplant)
* Life expectancy of at least 6 months without full VAD support

Exclusion Criteria:

* Age >75 years
* Exercise tolerance limited by factors other than heart failure
* Presence of intra-atrial thrombus
* Clinically significant right heart failure
* Serum creatinine >/= 2.5 mg/dl or any dialysis in previous 3 months
* Evidence of intrinsic hepatic disease
* Previous episode of resuscitated sudden death without subsequent treatment with AICD
* Subclavian artery stenosis
* Low platelet count, INR that cannot be corrected prior to implant or contraindication to anticoagulation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2007-06-29 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2018-01-29 (Actual)

PRIMARY OUTCOMES:
Safety - Adverse Events | 3 months
  Evaluation of the incidences of device failure or malfunction, adverse events associated with device use, surgical complications with device implant, and demonstration that the device provides adequate circulatory support in advanced HF patients.

SECONDARY OUTCOMES:
Change in hemodynamics | 3 months
  Evaluation of changes across time in hemodynamics, exercise tolerance, neurohormones, quality of life, functional capacity and ventricular function to determine the incidence of worsening HF in patients while supported by the CircuLite Synergy Device.

CONTACTS AND LOCATIONS:
Locations (11):
- UZ Leuven, Leuven, Belgium
- Germany (7):
  - German Heart Centre Berlin, Berlin
  - Heart Center Cologne University Hospital, Cologne
  - University Hospital Freiburg, Freiburg im Breisgau
  - Hannover Medical School, Hanover
  - Medical School Hannover, Hanover
  - Heart Centre University Leipzig, Leipzig
  - University Hospital Muenster, Münster
- Humanitas Clinical and Research Center, Milan, Italy
- National Institute of Cardiovascular Diseases Bratislava, Bratislava, Slovakia
- Harefield Hospital, Harefield, United Kingdom

REFERENCES:
- [Background] Morley D, Litwak K, Ferber P, Spence P, Dowling R, Meyns B, Griffith B, Burkhoff D. Hemodynamic effects of partial ventricular support in chronic heart failure: results of simulation validated with in vivo data. J Thorac Cardiovasc Surg. 2007 Jan;133(1):21-8. doi: 10.1016/j.jtcvs.2006.07.037. PMID 17198776
- [Derived] Meyns B, Klotz S, Simon A, Droogne W, Rega F, Griffith B, Dowling R, Zucker MJ, Burkhoff D. Proof of concept: hemodynamic response to long-term partial ventricular support with the synergy pocket micro-pump. J Am Coll Cardiol. 2009 Jun 30;54(1):79-86. doi: 10.1016/j.jacc.2009.04.023. PMID 19555845